CLINICAL TRIAL: NCT02803853
Title: Engaging Tribal Policy Makers to Sustain Improvements to the Food and Physical Activity Environments in American Indian Communities (OPREVENT2)
Brief Title: Engaging Tribal Policy Makers to Improve the Food and Physical Activity Environments in American Indian Communities
Acronym: OPREVENT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01HL122150-01A1 (NIH)
Record Dates: First submitted 2016-06-10; First posted 2016-06-17 (Estimated); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Obesity
Keywords: Native American; Obesity; Multi level; Policy; Schools; Worksite; Social Media; Food Store
MeSH Terms: conditions — Obesity | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): The intervention is a multi-level, multi-component intervention designed to increase access to and consumption of healthier foods in Native American Communities. Intervention components will occur at the policy level; food retail outlet level; neighborhood level- schools and worksites, and household level.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Similar to many community- based public health research programs, the control arm will not receive any intervention components during the initial intervention period. However, after all assessments are completed they will receive a 'delayed intervention' protocol, where the community receives the intervention elements as described in the intervention arm after assessment measures have been completed.

INTERVENTIONS:
Behavioral: Intervention — Intervention components will occur at the policy level (working with tribal leaders makers to sustain intervention components; food retail outlet level (working with grocery stores and owners to stock, promote, and sell healthier foods and beverages); neighborhood level (working with worksites and schools to deliver nutrition intervention sessions to youth and adults in intervention neighborhoods); household level (providing a social media program that provides parents and caregivers tips for healthier eating).
  Arms: Intervention

SUMMARY:
The overall objective of the study is to reduce adult obesity in participating American Indian (AI) communities and to improve understanding of the behavioral and environmental factors affecting obesity in these settings.

DETAILED DESCRIPTION:
The investigators plan to accomplish this objective by developing, implementing, and evaluating a randomized controlled trial of an intervention to improve diet and physical activity-related risk factors of obesity. A previous iteration of the intervention trial, called Obesity Prevention Research and Evaluation of InterVention Effectiveness in NaTive North Americans (OPREVENT) was implemented in five American Indian communities in Michigan and New Mexico. OPREVENT was a multi-level, multi-component intervention functioning at the community, institution, household, and individual levels and was implemented in schools, food stores, and worksites. Prior to OPREVENT, the research team has run multi-level interventions by working with schools and food stores in Native North American (NNA) communities1-6. For this new trial, named OPREVENT2, the research team will expand on the collective experience working on obesity prevention interventions in American Indian (AI) settings by developing complementary policy and social media components to support long-term sustainability of the OPREVENT intervention. OPREVENT2 will be implemented in six new AI communities.

ELIGIBILITY:
Inclusion Criteria:

* With the exception of the school intervention, which will only include teachers of grades 2-6 and students in grades 2-6 (ages 6-13), all community members will be included in the intervention.

Gender, Age and Locale

* The investigators will work with male and female schoolchildren and adults, aged 6-13 and 18-75 years who live in one of the participating tribal communities.

Exclusion Criteria:

* No adult community members will be excluded from the intervention as they are "passive" media and environmental changes, and available to everyone.

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 876 (Actual)
Dates: Start 2015-04; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | Up to 4 years
  The investigators will compare the mean change in BMI of participants living in intervention communities to those in the comparison communities, using data from the Adult Impact Questionnaire (AIQ). The investigators expect that the OPREVENT2 intervention will result in a 1.3 kg/m2 change in mean BMI, due to the multi-level, multi-component reinforcing design of this trial. These analyses will be adjusted for baseline value, participant and household (HH) covariates.

SECONDARY OUTCOMES:
The number of health-related policies under review | Up to 4 years
  The investigators will assess potential impact of the program by the increased number of health-related policies under review. The investigators will work to ensure that participating tribal leaders have the evidence base and tools to pass health-related policies and specifically policies that will work to support increased access to healthy foods and physical activity resources within communities.
Percent of time spent in sedentary activity and total activity counts | Up to 4 years
  The investigators will examine mean changes in participants' amount of time spent sitting, walking, doing moderate physical activity or doing vigorous physical activity (in the prior week) comparing pre- and post-intervention using the modified International Physical Activity Questionnaire-Short Form (IPAQ-SF). The investigators will use regression analysis to determine if participants' mean time spent inactive (i.e., sitting) decreases from pre- to post-intervention comparing intervention and control groups, adjusting for participant covariates and HH covariates.
Intake of fruits and vegetable servings,fiber, total energy and fat intake. | Up to 4 years
  Using a modified version of the Block Food Frequency Questionnaire (FFQ) the investigators will examine mean changes in participants' intake of fruit and vegetable servings (separately and aggregated), fiber intake, total energy and fat intake from pre- to post-intervention in intervention and control groups, using linear regression analysis, adjusting for baseline value of the outcome variable, participant covariates (e.g., age, sex) and household covariates (e.g., income, age and education).
Waist to hip ratio | Up to 4 years
  The investigators will compare the mean change in waist to hip ratio of participants living in intervention communities to those in the comparison communities, using data from the Adult Impact Questionnaire (AIQ). These analyses will be adjusted for baseline value, participant and household (HH) covariates.
Percent body fat | Up to 4 years
  The investigators will compare the mean change in % body fat of participants living in intervention communities to those in the comparison communities, using data from the Adult Impact Questionnaire (AIQ). These analyses will be adjusted for baseline value, participant and household (HH) covariates.

OTHER OUTCOMES:
Knowledge, self-efficacy, outcome expectations, and behavioral intentions | Up to 4 years
  The investigators will develop a series of scales to operationalize psychosocial factors (i.e., knowledge, self-efficacy, outcome expectations, and behavioral intentions).

CONTACTS AND LOCATIONS:
Overall Officials: Joel Gittelsohn, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed data sharing plan is intended to make study data as widely and freely available as possible, while safeguarding the privacy of participants, and protecting confidentiality. The data sharing plan includes additional stages of review and approval by the Navajo and Indian Health Services (IHS) Institutional Review Boards (IRBs). The investigators will strip the final dataset of personal identifiers prior to release for sharing. As even aggregated data may be perceived as stigmatizing, the investigators will make the data available to users under a data-sharing agreement that provides for: 1 initial approval of the data sharing request by the investigator, Navajo/IHS IRBs; 2 a commitment to not identifying participating communities without the express permission of that tribe's authorities; 3 a commitment to destroying or returning the data after analyses are completed; and 4 a commitment to having all manuscripts/documents approved by the Navajo/IHS IRBs prior to publication.

REFERENCES:
- [Derived] Redmond LC, Wensel CR, Estrade M, Fleischhacker SE, Poirer L, Jock BWI, Gittelsohn J. Dietary Outcomes of a Multilevel, Multicomponent, Cluster Randomized Obesity Intervention in 6 Native American Communities in the Upper Midwest and Southwest United States. Curr Dev Nutr. 2023 Feb 6;7(6):100043. doi: 10.1016/j.cdnut.2023.100043. eCollection 2023 Jun. PMID 37396963
- [Derived] Jock BWI, Maudrie T, Fleischhacker S, Porter KP, Gittelsohn J. Journey to Promoting Structural Change for Chronic Disease Prevention: Examining the Processes for Developing Policy, Systems, and Environmental Supports in Native American Nations. Curr Dev Nutr. 2022 Mar 16;6(3):nzab031. doi: 10.1093/cdn/nzab031. eCollection 2022 Mar. PMID 35310617
- [Derived] Gittelsohn J, Jock B, Redmond L, Fleischhacker S, Eckmann T, Bleich SN, Loh H, Ogburn E, Gadhoke P, Swartz J, Pardilla M, Caballero B. OPREVENT2: Design of a multi-institutional intervention for obesity control and prevention for American Indian adults. BMC Public Health. 2017 Jan 23;17(1):105. doi: 10.1186/s12889-017-4018-0. PMID 28114926